CLINICAL TRIAL: NCT06324851
Title: The Use of Drospirenone/Estetrol, Nomegestrol Acetate/Estradiol and Ethinylestradiol/Dienogest in Random Start Rapid Preparation of Endometrium Before Office Hysteroscopic Polypectomies: a Multicenter, Prospective, Randomized Study
Brief Title: The Use of Drospirenone/Estetrol, Nomegestrol Acetate/Estradiol and Ethinylestradiol/Dienogest in Random Start Rapid Endometrial Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, M.D., University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DROVZOEFFIPREP
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Polyp; Endometrial Diseases
Keywords: hysteroscopy; Endometrial preparation
MeSH Terms: conditions — Uterine Diseases | interventions — drospirenone and estetrol; nomegestrol acetate; Estradiol; Ethinyl Estradiol; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drospirenone/Estetrol (Experimental): Patients with endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Drospirenone/Estetrol at any time of the menstrual cycle
  Interventions: Drug: Drospirenone / Estetrol
- Nomegestrol Acetate/Estradiol (Experimental): Patients with endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Nomegestrol Acetate/Estradiol at any time of the menstrual cycle
  Interventions: Drug: Nomegestrol Acetate / Estradiol
- Ethinylestradiol/Dienogest (Experimental): Patients with endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Ethinylestradiol/Dienogest at any time of the menstrual cycle
  Interventions: Drug: Ethinylestradiol / Dienogest

INTERVENTIONS:
Drug: Drospirenone / Estetrol — Endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Drospirenone/Estetrol at any time of the menstrual cycle
  Arms: Drospirenone/Estetrol
Drug: Nomegestrol Acetate / Estradiol — Endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Nomegestrol Acetate/Estradiol at any time of the menstrual cycle
  Arms: Nomegestrol Acetate/Estradiol
Drug: Ethinylestradiol / Dienogest — Endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Ethinylestradiol/Dienogest at any time of the menstrual cycle
  Arms: Ethinylestradiol/Dienogest

SUMMARY:
The presence of a thin endometrium plays an important role in enabling the best conditions for hysteroscopic surgery. Recently, for this purpose, many studies have evaluated the effect of preoperative administration of a variety of drugs. We explored the efficacy of random started 14-day administration of Drospirenone/Estetrol or Nomegestrol Acetate/Estradiol or Ethinylestradiol/Dienogest, in rapid preparation of endometrium for hysteroscopic polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometrial polyps.

Exclusion Criteria:

* Patients with other endometrial pathologies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of endometrial preparation | 14th day of treatment
  Quality of endometrial preparation assessed visually intraoperatively by the surgeon using a visual analog scale from 0 to 5

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Andrea Etrusco, Palermo
  - Marco Monti, Rome